CLINICAL TRIAL: NCT01405911
Title: A Phase II, Randomized, Placebo-Controlled, Parallel-group, Double-Blind, Dose Response Finding Clinical Trial to Study the Efficacy and Safety of MK-0431/ONO-5435 in Japanese Subjects With Impaired Glucose Tolerance Who Have Inadequate Glycemic Control on Diet/Exercise Therapy
Brief Title: Dose Response Finding Study of MK-0431/ONO-5435 in Japanese Subjects With Impaired Glucose Tolerance (MK-0431-105)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-105; MK-0431-105 (Other: Merck Protocol Number)
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will take one tablet of placebo for sitagliptin 25 mg and one tablet of placebo for sitagliptin 50 mg orally once daily for 8 weeks.
  Interventions: Drug: Placebo for Sitagliptin 25 mg; Drug: Placebo for Sitagliptin 50 mg
- Sitagliptin 25 mg (Experimental): Participants will take one tablet of sitagliptin 25 mg and one tablet of placebo for sitagliptin 50 mg orally once daily for 8 weeks.
  Interventions: Drug: Placebo for Sitagliptin 50 mg; Drug: Sitagliptin 25 mg
- Sitagliptin 50 mg (Experimental): Participants will take one tablet of sitagliptin 50 mg and one tablet of placebo for sitagliptin 25 mg orally once daily for 8 weeks.
  Interventions: Drug: Placebo for Sitagliptin 25 mg; Drug: Sitagliptin 50 mg

INTERVENTIONS:
Drug: Placebo for Sitagliptin 25 mg — 1 tablet orally once daily before breakfast for 8 weeks
  Arms: Placebo; Sitagliptin 50 mg
Drug: Placebo for Sitagliptin 50 mg — 1 tablet orally once daily before breakfast for 8 weeks
  Arms: Placebo; Sitagliptin 25 mg
Drug: Sitagliptin 25 mg — 1 tablet orally once daily before breakfast for 8 weeks
  Other Names: MK-0431/ONO-5435
  Arms: Sitagliptin 25 mg
Drug: Sitagliptin 50 mg — 1 tablet orally once daily before breakfast for 8 weeks
  Other Names: MK-0431/ONO-5435
  Arms: Sitagliptin 50 mg

SUMMARY:
This study is being done to evaluate the safety, efficacy, and dose level of sitagliptin (MK-0431/ONO-5435) used once daily (qd) in Japanese participants with impaired glucose tolerance who have inadequate glycemic control using diet and exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance
* On diet/exercise therapy
* Unlikely to conceive
* Meets all of the following glycemic parameters: Hemoglobin A1c (Japan Diabetes Society value) <6.1%, Fasting Plasma Glucose <126 mg/dL, and 2-hr plasma glucose level in 75g oral glucose tolerance test ≥140 mg/dL and <200 mg/dL

Exclusion Criteria:

* History of diabetes mellitus
* Disease or condition of clear or likely glucose tolerance disorder
* Previously treated with a drug to prevent diabetes and/or any antihyperglycemic drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2011-08-16 (Actual); Primary Completion 2012-04-09 (Actual); Study Completion 2012-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Kaku K, Kadowaki T, Terauchi Y, Okamoto T, Sato A, Okuyama K, Arjona Ferreira JC, Goldstein BJ. Sitagliptin improves glycaemic excursion after a meal or after an oral glucose load in Japanese subjects with impaired glucose tolerance. Diabetes Obes Metab. 2015 Nov;17(11):1033-41. doi: 10.1111/dom.12507. Epub 2015 Jul 17. PMID 26094974

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received one tablet of placebo for sitagliptin 25 mg and one tablet of placebo for sitagliptin 50 mg orally once daily for 8 weeks.
- Sitagliptin 25 mg: Participants received one tablet of sitagliptin 25 mg and one tablet of placebo for sitagliptin 50 mg orally once daily for 8 weeks.
- Sitagliptin 50 mg: Participants received one tablet of sitagliptin 50 mg and one tablet of placebo for sitagliptin 25 mg orally once daily for 8 weeks.
Period: Overall Study
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg
Started | 83 | 82 | 77
Treated | 82 | 82 (1 participant received study drug but was discontinued due to pre-treatment lab AE.) | 77
Completed | 79 | 79 | 76
Not Completed | 4 | 3 | 1
Not completed — Pre-treatment lab AE | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg | Total
Number analyzed (Participants) | 83 | 82 | 77 | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (10.6) | 63.1 (9.5) | 61.9 (9.3) | 62.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 32 | 105
  Male | 48 | 44 | 45 | 137

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Glucose Total Area Under the Concentration Curve 0 to 2 Hours (AUC 0-2 Hrs) for Meal Tolerance Test (MTT) at Week 8
Description: Glucose total AUC 0-2 hours for MTT was measured at Baseline (Week 0) and at Week 8. After fasting for ≥10 hours, blood samples for glucose measurement were drawn at 0 minutes (at standard meal loading), 30 minutes, 60 minutes, 90 minutes, and 120 minutes. At Week 8, participants received study drug or placebo 30 minutes prior to consuming a standard meal.
Time Frame: Baseline (Week 0) and Week 8
Population: All participants, as randomized, who received at least one dose of study treatment and have a baseline measurement or post-randomization measurement for the analysis endpoint subsequent to study treatment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 82 | 82 | 77
Percent change | -2.42 [-4.48 to -0.31] | -9.52 [-11.43 to -7.57] | -11.49 [-13.40 to -9.55]
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin 25 mg; Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -7.11, 95% CI 2-sided [-9.85 to -4.36]
Statistical Analysis 2: Comparison: Placebo vs Sitagliptin 50 mg; Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -9.08, 95% CI 2-sided [-11.82 to -6.33]
Statistical Analysis 3: Comparison: Sitagliptin 25 mg vs Sitagliptin 50 mg; Test type: Other; p = 0.143, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -1.97, 95% CI 2-sided [-4.61 to 0.67]

2. Secondary Outcome: Percent Change From Baseline in Glucose Total Area Under the Concentration Curve 0 to 2 Hours (AUC 0-2 Hrs) for 75-gram Oral Glucose Tolerance Test (OGTT) at Week 7
Description: Glucose total AUC 0-2 hours for 75 g OGTT was measured at Baseline (Week -1) and at Week 7. After fasting for ≥10 hours, blood samples for glucose measurement were drawn at 0 minutes (at 75 g glucose loading), 30 minutes, 60 minutes, 90 minutes, and 120 minutes. At Week 7, participants received study drug or placebo 30 minutes prior to loading 75 g glucose solution.
Time Frame: Baseline (Week -1) and Week 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 82 | 82 | 77
Percent change | -3.68 [-6.66 to -0.60] | -21.38 [-23.81 to -18.87] | -20.09 [-22.61 to -17.48]
Statistical Analysis 1: Comparison: Placebo vs Sitagliptin 25 mg; Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -17.70, 95% CI 2-sided [-21.55 to -13.86]
Statistical Analysis 2: Comparison: Placebo vs Sitagliptin 50 mg; Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = -16.41, 95% CI 2-sided [-20.32 to -12.50]
Statistical Analysis 3: Comparison: Sitagliptin 25 mg vs Sitagliptin 50 mg; Test type: Other; p = 0.469, Constrained Longitudinal Data Analysis; Difference in Least Squares Means = 1.30, 95% CI 2-sided [-2.22 to 4.82]

3. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to 10 weeks
Population: All randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the actual study treatment they received. Due to a prescription error, one participant who was randomized to the placebo group took sitagliptin 50 mg.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 81 | 82 | 78
Percentage of participants | 30.9 | 34.1 | 41.0

4. Primary Outcome: Percentage of Participants Who Discontinued Treatment Due to an Adverse Event (AE)
Description: as for outcome 3
Time Frame: Up to 8 weeks
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg
Number analyzed (Participants) | 81 | 82 | 78
Percentage of participants | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Description: The analysis of safety data was based on all randomized participants who received at least one dose of study treatment. Participants were included in the treatment group corresponding to the actual study treatment they received. Due to a prescription error, one participant who was randomized to the placebo group took sitagliptin 50 mg.
Arm/Group | Placebo | Sitagliptin 25 mg | Sitagliptin 50 mg
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/82 | 0/78
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/82 | 0/78
Other Adverse Events (participants affected / at risk) | 13/81 | 14/82 | 11/78
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=81) | Sitagliptin 25 mg (N=82) | Sitagliptin 50 mg (N=78)
Nasopharyngitis (Infections and infestations) | 7 (7) | 9 (9) | 7 (7)
Hypoglycaemia (Metabolism and nutrition disorders) | 7 (7) | 5 (9) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.